CLINICAL TRIAL: NCT00868231
Title: Efficacy of Aclidinium Bromide Administered in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/23
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Antimuscarinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; BID protein, human; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Aclidinium 400 μg bid (Experimental): Aclidinium bromide 400 μg twice-daily by inhalation
  Interventions: Drug: Aclidinium bromide 400 μg bid
- Tiotropium 18 μg once-daily (Active Comparator): Tiotropium 18 μg once-daily by inhalation
  Interventions: Drug: Tiotropium 18 μg once-daily
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide 400 μg bid — Aclidinium bromide 400 μg twice-daily via inhalation by the Eklira Genuair® inhaler: 1 puff in the morning and evening for 15 days.
  Arms: Aclidinium 400 μg bid
Drug: Tiotropium 18 μg once-daily — Tiotropium 18 μg once-daily via inhalation by Handihaler® dry powder inhaler: 1 puff in the morning for 15 days.
  Arms: Tiotropium 18 μg once-daily
Drug: Placebo — Inhaled placebo: 1 puff in the morning (placebo to tiotropium) or in the morning and evening (placebo to aclidnium) for 15 days.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy, safety and tolerability of multiple doses of inhaled aclidinium bromide in moderate to severe COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients aged 40 with stable moderate to severe COPD (GOLD guidelines).
* Post-salbutamol (FEV1) < 80% and ≥ 30% of predicted normal value and Post-salbutamol FEV1/FVC < 70%.
* Current or ex smokers of 10 pack-years.

Exclusion Criteria:

* Patients with no history or current diagnosis of asthma.
* No evidence of an exacerbation within 6 weeks prior to the screening visit.
* No evidence of clinically significant respiratory and/or cardiovascular conditions or laboratory abnormalities.
* No contraindication to use of anticholinergic drugs such as known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (2):
- Germany (2):
  - Almirall Investigational Site #1, Berlin
  - Almirall Investigational Site #2, Großhansdorf

REFERENCES:
- [Derived] Fuhr R, Magnussen H, Sarem K, Llovera AR, Kirsten AM, Falques M, Caracta CF, Garcia Gil E. Efficacy of aclidinium bromide 400 mug twice daily compared with placebo and tiotropium in patients with moderate to severe COPD. Chest. 2012 Mar;141(3):745-752. doi: 10.1378/chest.11-0406. Epub 2011 Sep 8. PMID 21903737
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 sites in Germany. The first patient was screened in Mar 2009 and the last patient visit was in Jul 2009.
Pre-assignment Details: Eligible patients had at least a 5-day run-in period (and a maximum of 9 days) to assess patient's clinical stability.
Groups:
- Aclidinium 400 μg BID - Placebo - Tiotropium 18 μg: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium bromide from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
- Aclidinium 400 μg BID - Tiotropium 18 μg - Placebo: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium bromide from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
- Tiotropium 18 μg - Aclidinium 400 μg BID - Placebo: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium bromide from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
- Tiotropium 18 μg - Placebo - Aclidinium 400 μg BID: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the evening and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
- Placebo - Aclidinium 400 μg BID - Tiotropium 18 μg: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium bromide from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
- Placebo - Tiotropium 18 μg - Aclidinium 400 μg BID: The study consisted of 3 periods of 15 treatment days each separated by a washout period of 9 to 15 days.
  In treatment period 1, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 2, patients received 1 puff of placebo from the Eklira Genuair® inhaler and 1 puff of tiotropium from the Handihaler® inhaler in the morning and 1 puff of placebo from the Eklira Genuair® inhaler in the evening for 15 consecutive days.
  In treatment period 3, patients received 1 puff of aclidinium bromide from the Eklira Genuair® inhaler and 1 puff of placebo from the Handihaler® inhaler in the morning and 1 puff of aclidinium bromide from the Eklira Genuair® inhaler at in the evening for 15 consecutive days.
Period: Treatment Period 1
Arm/Group | Aclidinium 400 μg BID - Placebo - Tiotropium 18 μg | Aclidinium 400 μg BID - Tiotropium 18 μg - Placebo | Tiotropium 18 μg - Aclidinium 400 μg BID - Placebo | Tiotropium 18 μg - Placebo - Aclidinium 400 μg BID | Placebo - Aclidinium 400 μg BID - Tiotropium 18 μg | Placebo - Tiotropium 18 μg - Aclidinium 400 μg BID
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Aclidinium 400 μg BID - Placebo - Tiotropium 18 μg | Aclidinium 400 μg BID - Tiotropium 18 μg - Placebo | Tiotropium 18 μg - Aclidinium 400 μg BID - Placebo | Tiotropium 18 μg - Placebo - Aclidinium 400 μg BID | Placebo - Aclidinium 400 μg BID - Tiotropium 18 μg | Placebo - Tiotropium 18 μg - Aclidinium 400 μg BID
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 4 | 5 | 5 | 5 | 4 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Aclidinium 400 μg BID - Placebo - Tiotropium 18 μg | Aclidinium 400 μg BID - Tiotropium 18 μg - Placebo | Tiotropium 18 μg - Aclidinium 400 μg BID - Placebo | Tiotropium 18 μg - Placebo - Aclidinium 400 μg BID | Placebo - Aclidinium 400 μg BID - Tiotropium 18 μg | Placebo - Tiotropium 18 μg - Aclidinium 400 μg BID
Started | 4 | 5 | 5 | 5 | 4 | 5
Completed | 4 | 5 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All patients randomized into the crossover study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.9)
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Region of Enrollment [Number; unit: participants]
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-12 hr at Day 15 on Treatment.
Time Frame: Day 15
Population: Intention-to-treat (ITT) population; patients were included who took at least one dose of Investigational Medicinal Product and had at least a baseline and one post-dose value of FEV1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Aclidininum Bromide 400 μg Bid: Aclidinium bromide 400 μg twice-daily via inhalation
- Placebo: Placebo via inhalation
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 27
Liters | 0.236 (0.069) | 0.260 (0.070) | 0.015 (0.070)

2. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 12-24hr at Day 15 on Treatment
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 28 | 27
Liters | 0.174 (0.070) | 0.096 (0.070) | -0.032 (0.071)

3. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-24 hr at Day 15 on Treatment
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 28 | 27
Liters | 0.226 (0.063) | 0.178 (0.063) | -0.006 (0.063)

4. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC0-12) in Liters at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 30
Liters | 0.230 (0.040) | 0.178 (0.040) | 0.016 (0.040)

5. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 12-24 hr at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 27 | 29
Liters | 0.202 (0.051) | 0.101 (0.051) | -0.060 (0.050)

6. Secondary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-24 hr at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 29
Liters | 0.211 (0.044) | 0.138 (0.044) | -0.024 (0.044)

7. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 0-12 hr at Day 15 on Treatment
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 27
Liters | 0.297 (0.083) | 0.345 (0.083) | 0.009 (0.084)

8. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 12-24 hr at Day 15 on Treatment
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 28 | 27
Liters | 0.224 (0.074) | 0.087 (0.074) | -0.095 (0.075)

9. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 0-24 hr at Day 15 on Treatment
Time Frame: Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 28 | 27
Liters | 0.281 (0.078) | 0.219 (0.078) | -0.039 (0.078)

10. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 0-12 hr at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 30
Liters | 0.331 (0.064) | 0.289 (0.064) | 0.005 (0.063)

11. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 12-24 hr at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 28 | 27 | 29
Liters | 0.293 (0.072) | 0.150 (0.073) | -0.127 (0.072)

12. Secondary Outcome: Change From Baseline in Normalised Forced Vital Capacity (FVC) Area Under the Curve (AUC) 0-24 hr at Day 1 on Treatment
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 29 | 28 | 29
Liters | 0.310 (0.067) | 0.215 (0.067) | -0.051 (0.066)

ADVERSE EVENTS:
Arm/Group | Aclidininum Bromide 400 μg Bid | Tiotropium 18 μg Once-daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 1/30
Other Adverse Events (participants affected / at risk) | 2/29 | 0/28 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidininum Bromide 400 μg Bid (N=29) | Tiotropium 18 μg Once-daily (N=28) | Placebo (N=30)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidininum Bromide 400 μg Bid (N=29) | Tiotropium 18 μg Once-daily (N=28) | Placebo (N=30)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.